CLINICAL TRIAL: NCT05202379
Title: A Phase 1 Study in Healthy Participants to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single-Ascending and Multiple-Ascending Doses of the Influenza A Virus Replication Inhibitor CC-42344
Brief Title: CC-42344 Safety Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cocrystal Pharma, Inc. (Industry)
Collaborators: Cocrystal Pharma Australia Pty Ltd. (Unknown); Linear Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: CC-42344-P1-001
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Influenza A
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 4 cohorts for SAD, with food cohort; 5 cohorts for MAD; 6 active and 2 placebo per cohort; 6 additional active in food cohort
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: active and placebo capsules identical visually.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- SAD cohort 1A (Experimental): first dose level with 6 active and 2 placebo healthy participants
  Interventions: Drug: CC-42344; Drug: Placebo
- SAD cohort 1B (Experimental): second dose level with 6 active and 2 placebo healthy participants
  Interventions: Drug: CC-42344; Drug: Placebo
- SAD cohort 1C (Experimental): third dose level with 12 active and 2 placebo healthy participants; food-effect cohort
  Interventions: Drug: CC-42344; Drug: Placebo
- SAD cohort 1D (Experimental): fourth dose level with 6 active and 2 placebo healthy participants
  Interventions: Drug: CC-42344; Drug: Placebo
- MAD cohort 2A (Experimental): first dose level with 6 active and 2 placebo healthy participants dose x 14 days
  Interventions: Drug: CC-42344; Drug: Placebo
- MAD cohort 2B (Experimental): second dose level with 6 active and 2 placebo healthy participants dose x 14 days
  Interventions: Drug: CC-42344; Drug: Placebo
- MAD cohort 2C (Experimental): third dose level with 6 active and 2 placebo healthy participants dose x 14 days
  Interventions: Drug: CC-42344; Drug: Placebo
- MAD cohort 2D (Experimental): forth dose level with 6 active and 2 placebo healthy participants dose x 5 days
  Interventions: Drug: CC-42344; Drug: Placebo
- MAD cohort 2E (Experimental): forth dose level with 6 active and 2 placebo healthy participants dose x 5 days
  Interventions: Drug: CC-42344; Drug: Placebo

INTERVENTIONS:
Drug: CC-42344 — CC-42344 capsules
  Other Names: Active
Drug: Placebo — Placebo capsules

SUMMARY:
CC-42344 Phase 1 study with single-ascending dose (SAD) and multiple-ascending dose (MAD) parts.

DETAILED DESCRIPTION:
This study is testing the safety, tolerability, and pharmacokinetics (PK, the amount of study drug in the blood) of a new drug called CC-42344.Up to 78 healthy men or women aged between 18-55 are planned to be enrolled in this study in two parts.

Part 1 will involve a single-ascending (increasing) dose (SAD) where 32 participants (4 groups of 8) will be assigned randomly to receive a single oral dose of the study drug or placebo. The placebo will look the same as the study drug but will not contain any medicine. An additional 6 participants will receive a single oral dose of CC-42344 to help further understand the effect of food on the uptake of the drug.

Part 2: will involve a multiple-ascending dose (MAD) where 40 participants (5 groups of 8) will be randomized to receive an oral dose of study drug or placebo given once a day for 14 days, once a day for 5 days, or twice a day for 5 days. The placebo will look the same as the study drug but will not contain any medicine.

ELIGIBILITY:
Inclusion Criteria (main):

* Healthy males or healthy, non-pregnant, non-lactating females
* Body weight of at least 50 kg
* Body mass index between ≥18.0 and ≤32.0 kg/m2
* Good state of health (mentally and physically)
* Negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test, if required and per site policy

Exclusion Criteria (main):

* Have received any investigational drug in a clinical research study within the previous 30 days before screening
* Have received any vaccine within 7 days prior to randomization
* History of any drug or alcohol abuse in the past 2 years
* Females of childbearing potential who are pregnant or lactating or planning to become pregnant during the study
* Clinically significant abnormal biochemistry, hematology, coagulation, or urinalysis as judged by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
treatment emergent adverse events | Day 1 to 7 days after last dose
  number of participants with treatment-emergent adverse events
laboratory abnormalities | Day 1 to 7 days after last dose
  number of participants with clinically significant laboratory abnormalities
vital signs | Day 1 to 7 days after last dose
  number of participants with clinically significant changes from baseline in vital signs
ECG | Day 1 to 7 days after last dose
  number of participants with clinically significant changes from baseline in ECGs

SECONDARY OUTCOMES:
maximum plasma concentration | Day 1 to 7 days after last dose
  measurement of maximum plasma concentration (Cmax)
time of maximum plasma concentration | Day 1 to 7 days after last dose
  measurement of time of maximum plasma concentration (Tmax)
area under the plasma concentration-time curve | Day 1 to 7 days after last dose
  measurement of area under the plasma concentration-time curve (AUC)
elimination rate constant | Day 1 to 7 days after last dose
  measurement of elimination rate constant
terminal elimination half-life | Day 1 to 7 days after last dose
  measurement of terminal elimination half-life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Salman, MD, Principal Investigator — Linear Clinical Research
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No